CLINICAL TRIAL: NCT06549257
Title: A Phase Ib Open Label Clinical Trial of the Safety, Immunogenicity and ex Vivo Efficacy of Two Candidate Malaria Transmission Blocking Vaccines, Pfs25-IMX313 and Pfs45/48 Administered Alone and in Combination, in Matrix-M Adjuvant in Healthy Adults, Adolescents and Young Children in Burkina Faso
Brief Title: Assessing the Safety, Immunogenicity and Ex-vivo Efficacy of Two Candidate Malaria Transmission Blocking Vaccines, Pfs25-IMX313 and Pfs45/48 Administered Alone and in Combination, in Matrix-M Adjuvant
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC099
Record Dates: First submitted 2024-03-12; First posted 2024-08-12 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-08

CONDITIONS: Plasmodium Falciparum Malaria
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - Pfs25-IMX313 (Experimental): Vaccination with three doses of Pfs25-IMX313 10ug in 50ug Matrix M.
  Interventions: Biological: Pfs25-IMX313, Pfs48/45
- Group 2 - Pfs48/45 (Experimental): Vaccination with three doses of Pfs48/45 10ug in 50ug Matrix M.
  Interventions: Biological: Pfs25-IMX313, Pfs48/45
- Group 3 - Pfs25-IMX313 and Pfs48/45 (Experimental): Vaccination with three doses of Pfs25-IMX313 10ug in 50ug Matrix M and vaccination with three doses of Pfs48/45 10ug in 50ug Matrix M.
  Interventions: Biological: Pfs25-IMX313, Pfs48/45

INTERVENTIONS:
Biological: Pfs25-IMX313, Pfs48/45 — Two soluble protein vaccines.

SUMMARY:
Assessing the safety, immunogenicity and ex-vivo efficacy of two transmission blocking vaccines (Pfs25-IMX313 in Matrix M and Pfs48/45 in Matrix M alone and co-administered) in Burkina Faso, in 18-45 years, 12-17 years and 05-11 year olds.

ELIGIBILITY:
Inclusion Criteria:

All volunteers must satisfy all the following criteria to be eligible for the study

* Healthy adults, adolescents and children based on medical history, physical examination and baseline blood tests
* Age: 5-45 years of age at the time of enrollment (i.e. up to the day before their 46th birthday).
* Signed informed consent/thumb-printed and witnessed informed consent obtained from the parent(s)/guardian(s) of the participant to join the trial (if under the age of 18). For participants aged 18 and above, signed informed consent/thumb-printed of the participant.
* Signed informed assent/thumb-printed and witnessed assent obtained from participants (for age group 12-17 years old only).
* The investigator believes that the participant and their parents/guardians (if participant aged under 18) can and will comply with the requirements of the protocol.
* The participant is a permanent resident of the study area and likely to remain a resident for the duration of the trial.
* Agreement to refrain from blood donation for the duration of the study
* Female participants of childbearing potential (WOCBP) must agree to avoid pregnancy during the duration of the study and practice continuous effective contraception if sexually active.

Acceptable forms of contraception for female volunteers of childbearing potential include:

* Established use of oral, injected or implanted hormonal methods of contraception.
* Placement of an intrauterine device (IUD) or intrauterine system (IUS).
* Total abdominal hysterectomy.
* Sex abstinence/not sexually active

Exclusion Criteria

* The volunteer has previously received a malaria vaccine.
* The volunteer is enrolled in another malaria intervention trial.
* The volunteer is currently participating in another clinical trial if likely to affect data interpretation of either trial.
* The volunteer has a history of allergic disease or reactions likely to be exacerbated by any component of the study vaccines.
* The volunteer has a history of allergic reactions, significant IgE-mediated events or anaphylaxis to previous immunisations.
* The volunteer has anaemia associated with clinical signs of decompensation, or a haemoglobin of ≤ 7.4 g/dL
* The volunteer has been administered immunoglobulins and/or any blood products including blood transfusion within the three months preceding the planned administration of the vaccine candidate.
* Receipt of a vaccine 30 days prior to study vaccine administration or planning to receive one within 30 days after administration of any of the doses of the study vaccine.
* The volunteer has malnutrition requiring hospital admission.
* The volunteer has an acute or chronic, clinically significant pulmonary, cardiovascular, gastrointestinal, endocrine, neurological, skin, hepatic or renal functional abnormality, as determined by medical history, physical examination or laboratory tests
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Pregnancy, lactation or intention to become pregnant during the study.
* Hepatitis B surface antigen (HBsAg) detected in serum.
* Antibodies to HCV (HCV-Ab) detected in serum.
* Any other significant disease, disorder, or finding which, in the opinion of the investigator, may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

The following criteria should be checked during the study, prior to each vaccination:

• Any significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To assess safety and reactogenicity of Pfs25-IMX313-Matrix-M, Pfs48/45-Matrix M administered alone or in combination, in healthy Burkinabé adolescents and children naturally exposed to malaria. | Through study completion, an average of 8 months from enrollment
  Occurrence of solicited local and systemic reactogenicity signs and symptoms after each vaccination during a 7-day surveillance period (day of vaccination and days 1, 2, 3, 5 and 6 after vaccination).
  * Occurrence of unsolicited adverse events (AE) including safety laboratory measures for 28 days following each vaccination
  * Occurrence of serious adverse events (SAEs) during the whole study duration
  * Occurrence of AEs of special interest (AESIs) during the whole study duration

SECONDARY OUTCOMES:
To determine the Pfs25 and Pfs48/45 humoral immune response | Through study completion, an average of 8 months from enrolment
  Pfs25 and Pfs48/45 antibody levels elicited by Pfs25IMX313-Matrix-M and Pfs48/45 in Matrix-M as measured by ELISA at Days 0, 14, 28, 42, 56, 72, 140, 236
To determine the ex-vivo functional transmission blocking activity of Pfs25 and Pfs48/45 administered alone and in combination | Through study completion, an average of 8 months from enrolment
  Standard membrane feeding assays (SMFA) and direct membrane feeding assays (DMFA) at Days 0, 14, 28, 42, 56, 72, 140, 236, reported as a percentage of transmission reducing activity compared to controls (% TRA).

CONTACTS AND LOCATIONS:
Overall Officials: Paola Cicconi, PhD, Principal Investigator — University of Oxford

IPD SHARING:
Plan to Share IPD: Yes
Publication of the trial results via a peer reviewed journal
Time Frame: Approximately one year following the end of the trial